CLINICAL TRIAL: NCT06171594
Title: The Effect of Chlorhexidine on the Oral Microbiome, Salivary Pellicle Proteins and Vascular Function in Individuals With Dental Erosion
Brief Title: The Effect of Chlorhexidine on the Oral Microbiome and Saliva in Dental Erosion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Portsmouth (Other)
Responsible Party: Principal Investigator, Ant Shepherd, Dr Ant Shepherd - associate professor in clinical exercise physiology, University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 333173
Record Dates: First submitted 2023-11-09; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-11

CONDITIONS: Dental Erosion
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active chlorhexidine (Active Comparator): Arm Description 2: Antibacterial CHX Mouthwash Arm
  This arm involves participants who have been randomly assigned to receive an antibacterial CHX mouthwash containing 0.2% CHX (Corsodyl Mint, GlaxoSmithKline, UK). Similar to Arm 1, the intervention period spans seven days, during which participants will rinse their mouth with 10 mL of antibacterial CHX mouthwash twice daily. The active CHX mouthwash and the placebo mouthwash are indistinguishable in taste, appearance, color, texture, and smell. Participants in this arm will follow the rinse regimen for 7 days, taking the final tube the morning before their next visit (Visit 2 - 8). After the completion of Visit 8, each participant will undergo a washout period of 12 weeks before starting the 7-day reverse order of the given product administration as part of the crossover design.
  Interventions: Combination Product: Chlorhexidine mouthwash
- Placebo Chlorhexidine (Placebo Comparator): Arm Description 1: Placebo CHX Mouthwash Arm
  This arm involves participants who have been randomly assigned to receive a placebo CHX mouthwash. The intervention period spans seven days, during which participants in this arm will rinse their mouth with 10 mL of CHX placebo mouthwash (ultrapure mint-flavoured water) twice daily. The placebo mouthwash is designed to be identical in taste, appearance, colour, texture, and smell to the active mouthwash, ensuring blinding during the study. Participants in this arm will follow the rinse regimen for 7 days, taking the final tube the morning before their next visit (Visit 2 - 8). After the completion of Visit 8, each participant will undergo a washout period of 12 weeks before starting the 7-day reverse order of the given product administration as part of the crossover design.
  Interventions: Combination Product: Chlorhexidine mouthwash

INTERVENTIONS:
Combination Product: Chlorhexidine mouthwash — The proposed study is part of a PhD educational project and will be a double blind, randomised design, crossover trial for the effect of Chlorhexidine (CHX) mouthwash on healthy control and people with dental erosion (PwDE). This study aims to explore mouthwash's effect on oral microbiome recovery in WMS and salivary pellicle and its impact on blood pressure and arterial stiffness in healthy controls PwDE

SUMMARY:
Dental erosion happens when the teeth lose some of their parts because of acid from the things people eat and/or drink or even from stomach. It can make teeth hurt and become sensitive. The mouth has a protective shield called salivary pellicle that helps, and there are some special bacteria called Nitrate-reducing bacteria (NRB) that can be good for the mouth and heart. Eating some fruits and vegetables or drinking beetroot can make these bacteria thrive, which might help the heart and blood pressure. This study wants to see how administering chlorhexidine mouthwash affects the good bacteria in the mouth for people with healthy teeth and those with erosion. This study aims to find out if this mouthwash can change the saliva and bacteria in the mouth for the better, in people with both healthy teeth and those with dental erosion.

The proposed study is part of a PhD educational project and will be a double blind, randomised design, crossover trial for the effect of Chlorhexidine (CHX) mouthwash on healthy control and people with dental erosion (PwDE). This study aims to explore mouthwash's effect on oral microbiome recovery in WMS and salivary pellicle and its impact on blood pressure and arterial stiffness in healthy controls PwDE

DETAILED DESCRIPTION:
Upon consent being granted, several samples and measurements will be collected from the participant during this research study spanning over 15 visits. The proposed study will be a double blind, randomised design, crossover trial for the effect of CHX mouthwash on healthy control and PwDE. Two groups of participants are required for this study [healthy (n=12) and PwDE (n=12) groups] from volunteer participants from the university of Portsmouth (UoP) who have no signs of or reported medical problems (detailed protocol of recruitment attached). Based on power calculation, 14 individuals will be recruited for each group (healthy and PwDE groups) to account for a 14% drop-out rate.

Participants will be approached to volunteer for the study by the chief investigator and PhD researcher through word of mouth, emails via departmental staff lists, University of Portsmouth Dental Academy (UPDA) updates newsletter, UPDA department meetings and presentations about the study during the UPDA's journal club event. A participant information sheet (PIS) and consent form (see attached forms) will be distributed either via email or by handing out hard copies to those wishing to partake in the research. Participants who have returned their completed consent form will be invited to come to UPDA for further assessment of suitability (visit 1).

The participants who has agreed to take part in this research will be invited to attend the University of Portsmouth Dental Academy, Beatty Building (UPDA) for fifteen consecutive visits. They will be invited to attend the UPDA's dental clinics for their first visit for clinical screening and baseline sampling then for their consecutive sampling visits (14 visits) to attend Spinnaker Building, School of Sport, Health & Exercise Science, University of Portsmouth (SbUoP) for further sampling.

Visit 1 (30 minutes-1 hour): This visit will include clinical screening, consent and baseline samples taken and will take place at UPDA dental clinics. The mouths of participants will be screened for suitability to fit in either of the groups (healthy or dental erosion groups) depending on the presence or absence of dental erosion in their teeth. A BEWE will be used to screen as whether participants have erosion or not. It is a simple, reproducible and convenient scoring system that can be used for recording clinical findings of dental erosion. If BEWE score is greater than 8 per extant cumulative score and one score 3 in at least one sextant then this means the participant's mouth shows evidence of dental erosion. If a participant is found to be suitable based upon inclusion/exclusion criteria (see attached detailed protocol), they will be invited to attend further appointments.

A medical history, dental history and two further questionnaires (Diet Questionnaire and Reflux Disease Questionnaire) will be completed to ensure that they are suitable for this research study.

After the oral assessment and completing all forms and questionnaires, participants will be assigned to two groups of participants [healthy (n=12) and dental erosion (n=12) groups]. Within each group, the twelve participants will be randomly and blindly assigned to further two subgroups by an independent researcher to receive one of the mouthwash treatments [[placebo CHX group (n=6) and antibacterial CHX mouthwash group (n=6)] as can be seen in the attached protocol. In the same visit, they will then be invited to come to the science laboratory (Beatty Building, UPDA) for several sample collections. As described in the protocol and participant information sheet, these will include measuring participants' blood pressure and brachial artery endothelium-dependent function. Next, venous blood will be collected via venepuncture from the forearm in 4 mL aliquots. After that, saliva and salivary pellicle from teeth and tongue will be collected.

Then each participant from each subgroup will either receive 14 tubes containing 10 mL CHX placebo mouthwash (ultrapure mint-flavoured water) or another 14 tubes containing 10 ml antibacterial mouthwash containing 0.2% CHX (Corsodyl Mint, GlaxoSmithKline, UK) depending on the randomisation process. Both versions of the mouthwash will be identical in taste, appearance, colour, texture, and smell using plain, identical bottles for both solutions. They will be instructed to administer each product in a reverse order which will thoroughly be explained by a member of our research team during this visit (visit 1). Specifically, participants will be instructed to rinse their mouth with the selected mouthwash for 1 minute, twice a day for 7 days taking the final tube the morning before their next visit (visit2). For study standardisation, participants will also be given a standardised toothpaste to use throughout the duration of the study.

Visit 2 - 8 (30-40 minutes per visit):

Seven days after visit 1, participants will be invited to return to the (SbUoP) for visit 2, between 9AM-12PM, with the final dose being administered 2 hours prior to their scheduled appointment time. Upon arrival, blood pressure of the brachial artery (forearm) will be measured following 30 minutes of seated rest in a quiet room using an automated sphygmomanometer. A total of five successive measurements will be taken, with 1-minute rest between readings, with the mean of the final three measurements to be recorded. The mean of the systolic (SBP), diastolic (DBP) and mean arterial pressure (MAP) measurements will also be recorded. Endothelial function test and brachial artery endothelium-dependent function will be measured as described below in the analysis section. Next, venous blood will be collected via venepuncture from the forearm in 4 mL aliquots as described in the analysis section. Finally, WMS, AEP and tongue SP samples will then be collected as described in the detailed sample collection section below.

All participants will then be invited to come to the (SbUoP) for further six visits in which same samples and measurements will be collected.

Upon completion of final sample collections (visit 8), each participant from each group [healthy control (n=6) and PwDE(n=6)] will receive the reverse order of the product they had received in visit 1 (cross over) to be used after a washout period of 12-weeks. Each participant will either receive 14 tubes containing 10 mL CHX placebo mouthwash (ultrapure mint-flavoured water) or another 14 tubes containing 10 ml antibacterial mouthwash containing 0.2% CHX (Corsodyl Mint, GlaxoSmithKline, UK) in the reverse order (crossover design) depending on what they have had before the washout period (visit1) as seen in figure1.

Washout and Reverse treatment:

After visit 8, participants will be instructed to carry out a washout period of 12-weeks before starting the 7-day reverse order of the given product administration as above. Specifically, the 6 participants from each group [healthy (n=12) and PwDE (n=12)] who had administered placebo CHX mouthwash before visit 2 will be given same amount of antibacterial mouthwash containing 0.2% CHX (Corsodyl Mint, GlaxoSmithKline, UK) to be administered in the same conditions as explained above (1 min, twice daily for 7 days) with the final tube taken the morning before their next visit (visit 9). The other 6 individuals will be instructed to administer the placebo CHX in the reverse order (crossover) of their 5 counterparts during visit 2 as shown in figure 1, twice daily, with the final tube to be taken the morning before visit 9.

Visit 9 - 15 (30-40 minutes per visit):

Visit 9 will take place after the 12-week washout period followed by seven days of administering the reverse product as seen in figure 1. Participants will be invited to return to the (SbUoP), between 9AM-12PM, with the final dose being taken 2 hours prior to their scheduled appointment time (visit 9). Upon arrival, same sample and measurements will be repeated as visits (2-8). Upon completion of final sample collections (visit 15), this will be the end of volunteer participation.

ELIGIBILITY:
Inclusion Criteria:

- Eligibility Criteria A) Healthy volunteers Group

Inclusion Criteria:

1. Be aged 18 to 75 years inclusive
2. Have a minimum of 20 natural uncrowned teeth (excluding 3rd molars) present
3. Give written informed consent
4. Be in good general health and oral health (without active caries lesions, gingivitis, periodontitis.
5. No diseases of the soft or hard tissues of the oral cavity
6. No other oral condition affecting the composition of the oral fluids and presented normal salivary flow (stimulated salivary flow >1 mL/min, unstimulated salivary flow > 0.25 mL/min; salivary pH > 6)
7. Show no evidence of dental erosion or/and active dental caries (with BEWE score ≤8 per extant cumulative score per patient and no clinically visible decayed teeth) B) Dental erosion group Inclusion Criteria

1. Same as above of healthy volunteers (1-6). 2. Show evidence of dental erosion (with BEWE score > 8 per extant cumulative score per patient and one score 3 in a sextant. BEWE is a simple, reproducible and convenient scoring system that can be used with the diagnostic criteria for recording clinical findings and examining dental hard tissues other than for caries, guiding the management of erosive tooth wear.

Exclusion Criteria:

-

Exclusion Criteria for both groups:

1. Smokers, using mouthwash or tongue scrapes
2. Presenting conditions associated with vomiting (e.g. anorexia or bulimia), bruxism and Gastro-oesophageal reflux disease (GORD)
3. Occupations associated with increased risk of erosion, such as swimmers and battery, charging and galvanizing workers.
4. Wearing orthodontic appliances
5. Use of antibiotics three (3) months prior to or during this study
6. Use of any over the counter medications other than analgesics
7. Pregnant or breastfeeding
8. Participation in another clinical study in the month preceding this study
9. Medical condition which requires pre-medication prior to dental visits/procedures.
10. Participants who have eaten/had anything to drink up to two hours before providing a sample (Two hours prior to the trial, participants will be instructed to eat a self-selected light meal and drink 500 ml of water. No other food or fluid will be allowed thereafter)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Identification of salivary proteins via SDS-PAGE Electrophoresis: | Baseline (day -7), post each intervention (i.e. mouthwash and placebo) on days 0,1,3,7,14,21,28
  SDS-PAGE will be used to identify salivary proteins in saliva and pellicle samples and any potential changes in protein bands at a variety of conditions.
Identification of salivary proteins via Proteomics analysis: | Baseline (day -7), post each intervention (i.e. mouthwash and placebo) on days 0,1,3,7,14,21,28
  will identify a number of salivary proteins in saliva and pellicle samples including prolactin inducible protein (PIP) and zinc-alpha-2 glycoprotein (ZAG)
Microbiome diversity using DNA extraction and 16s ribosomal RNA analysis | Baseline (day -7), post each intervention (i.e. mouthwash and placebo) on days 0,1,3,7,14,21,28
  Saliva and pellicle samples will be used to isolate bacterial DNA which will be quantified using a fluorometric method Results from the DNA sequencing will be directly compared between those individuals classified as showing dental erosion and those healthy participants.

SECONDARY OUTCOMES:
Blood pressure measurement: | Baseline (day -7), post each intervention (i.e. mouthwash and placebo) on days 0,1,3,7,14,21,28
  Blood pressure of the brachial artery will be measured following 30 minutes of seated rest in a quiet room using an automated sphygmomanometer. A total of five successive measurements will be taken, with 1-minute rest between readings, with the mean of the final three measurements will be recorded. The mean of the systolic (SBP), diastolic (DBP) and mean arterial pressure (MAP) measurements will be recorded.
Endothelial function test (Iontophoresis) of brachial artery: | Baseline (day -7), post each intervention (i.e. mouthwash and placebo) on days 0,1,3,7,14,21,28
  Iontophoresis will permit the transdermal delivery of Acetylcholine (Ach) and sodium nitroprusside (SNP) to the volar aspect of the right forearm. These chemicals will be introduced through a process called Iontophoresis. Iontophoresis is a unique test where we use a gentle electrical charge to help specific substances get into your skin. This method is beneficial for carefully delivering therapeutic agents through skin or for diagnostic reasons.
Flow-mediated dilation (FMD) of brachial artery: | Baseline (day -7), post each intervention (i.e. mouthwash and placebo) on days 0,1,3,7,14,21,28
  Brachial artery endothelium-dependent function will be measured using the FMD technique as previously described. FMD represents an endothelium-dependent, largely NO-mediated dilatation of conduit arteries in response to an imposed increase in blood flow and shear stress. A high-resolution ultrasound machine will be used to image the brachial artery in the distal third of the upper arm.
Nitrate and nitrite in saliva, plasma via Ozone-based chemiluminescence | Baseline (day -7), post each intervention (i.e. mouthwash and placebo) on days 0,1,3,7,14,21,28
  Blood samples:
  Venous blood will be collected and analysed for NO3- and NO2- content
  Saliva samples:
  The WMS will be collected and analysed for NO3- and NO2- content
Oxidative stress markers and redox-related molecules via ELISA: | Baseline (day -7), post each intervention (i.e. mouthwash and placebo) on days 0,1,3,7,14,21,28
  ELISA will be used to identify some common Oxidative stress markers and redox-related molecules such as 3-NO-Tyr in saliva and blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth Academy, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan